CLINICAL TRIAL: NCT04699604
Title: A Histamine Pharmacodynamic Biomarker to Guide Treatment in Pediatric Asthma
Brief Title: A Histamine Pharmacodynamic Biomarker to Guide Treatment in Pediatric Asthma (HAS3)
Acronym: HAS3
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Bridgette Jones (Other)
Collaborators: Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD) (NIH)
Responsible Party: Sponsor-Investigator, Bridgette Jones, Medical Director and Associate Professor of Pediatrics, Children's Mercy Hospital Kansas City
Organization: Children's Mercy Hospital Kansas City (Other)
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Treatment
Other Study IDs: STUDY00001262; 5R01HD100545-05 (NIH)
Record Dates: First submitted 2020-12-30; First posted 2021-01-07 (Actual); Last update posted 2025-04-08 (Actual); Status verified 2025-04

CONDITIONS: Allergic Asthma
MeSH Terms: interventions — levocetirizine

STUDY DESIGN:
Intervention Model Description: Randomized, double-blind, placebo-controlled, crossover study
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Identity of the study article will be known only by the investigational pharmacist charged with dispensing the product and the research coordinator responsible for administering the study articles and obtaining timed blood specimens associated with pharmacokinetic and pharmacodynamic study objectives. Blinding of the principal investigator and co-investigators will be safeguarded by blinding the identity of the study articles (LTZ 0.5 mg/ml oral solution or placebo solution similar in color, flavoring and consistency) and preventing access to specific source documents that will be used for recording of collected blood samples until the time of data analysis.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Levocetirizine (LTZ) (Active Comparator): Participants will take Levocetirizine dihydrochloride/ Xyzal® (UCB, Inc.) immediate release oral solution 2.5mg/5ml (2.5mg in children 6-11 years of age; 5mg in children >11 years per recommended doses) in addition to their current asthma regimen.
  Interventions: Drug: Levocetirizine Dihydrochloride
- Placebo (Placebo Comparator): Participants will take a placebo solution previously developed by the Children's Mercy Investigational Pharmacy to match the color, flavor, and consistency of the active drug in addition to their current asthma regimen.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Levocetirizine Dihydrochloride — At the end of the HILD assessment participants will be randomized to Levocetirizine Dihydrochloride or placebo. Children will be randomized by an investigational pharmacist to add-on either Levocetirizine dihydrochloride/ Xyzal® (UCB, Inc.) immediate release oral solution 2.5mg/5ml (2.5mg in children 6-11 years of age; 5mg in children >11 years per recommended doses) or placebo to their current asthma regimen.
  Other Names: Xyzal
  Arms: Levocetirizine (LTZ)
Drug: Placebo — Placebo
  Arms: Placebo

SUMMARY:
This is a randomized, double-blind, placebo-controlled, crossover study comparing asthma control post treatment in African American/Black and Caucasian/White children in both hyper and hypo responsive HILD (Histamine Lontophoresis with Laser Doppler monitoring) phenotypes with uncontrolled persistent allergic asthma using Levocetirizine (LTZ) vs placebo.

DETAILED DESCRIPTION:
The investigator hypothesizes that children with a hyper-responsive HILD (Histamine Lontophoresis with Laser Doppler monitoring) response type are more likely to have improved asthma control after the addition of the antihistamine LTZ (Levocetirizine) to standard asthma regimen in comparison to children with hypo-responsive HILD type. This study will provide a model for a functional biomarker to inform decision making for therapeutics in children. This work is novel in testing and validating a biomarker accurately and predicting response to asthma treatment in children. This work is significant because it has the potential to alter the current treatment paradigms for children with asthma where response to treatment is predicted a priority. The proposed research will be immediately relevant by expanding knowledge in the field of asthma therapeutics by linking biologically and mechanistically based approaches to an effective and inexpensive treatment for asthma. The primary objective is to determine HILD prediction of therapeutic response in males and females 6-17 years old who identify as African American/Black and Caucasian/White to an antihistamine among children with allergic asthma, and the secondary objective is to develop a robust predictive model of therapeutic response to an antihistamine among children with allergic asthma. There will be 300 participants for approximately 17 weeks.

The primary outcome measure of therapeutic response to antihistamine will be determined by change in asthma control as guidelines recognize asthma control as a major goal of therapy. Asthma control will be determined based on the Asthma Control Test (ACT®) (children ≥ 12 years of age) or the Child-Asthma Control Test (C-ACT®) (children <12 years of age), validated measures to assess asthma control in children. Children with an ACT or C-ACT score <19 will be classified as having uncontrolled asthma. Assessments will occur at screening, visit 2, 3 and 4 (6 weeks after the participant is started on drug/placebo.) The secondary measures will include assessment of asthma impairment, risk, and quality of life. These assessments will occur at baseline/pre-dose, 6 weeks after starting drug/placebo, and 6 weeks after drug/placebo for both the LTZ and placebo arms.

The study team is utilizing HILD a surrogate marker of histamine response and will determine if HILD can predict which participants have improvement in asthma control after treatment with Levocetirizine.

ELIGIBILITY:
Inclusion Criteria:

1. A diagnosis of asthma based on physician diagnosis
2. A diagnosis of uncontrolled asthma based on Asthma Control Test (ACT) score within the last 3 months or at screening
3. Evidence of allergic sensitization based on allergy skin test or allergy blood test results
4. Individuals who are currently being treated with asthma guideline-based therapy
5. Males and females 6 through 17 years of age at time of enrollment
6. Willing to provide written permission/assent to participate
7. Children who self-identify as African American/black (identify both 1st degree (parents) and 2nd degree relatives (grandparents) as African American) or Caucasian/white (self-report of 1st and 2nd degree relatives as Caucasian)

Exclusion Criteria:

1. For females, positive pregnancy test (by urinary hCG) or lactation at the time of the study
2. Any other chronic disease states such as history of premature lung disease, bronchiectasis, cystic fibrosis, or any chronic lung disease other than asthma.
3. Chronic abnormal conditions of the liver or kidney, immunologic/hematologic, or neoplastic disease as determined by the PI (the following questions will be asked at initial screening to identify children with potential abnormal kidney function:

   Have you ever been diagnosed with chronic kidney disease?; Have you ever had to be on dialysis or take medications for chronic kidney disease?)
4. Inability or unwillingness to have blood drawn as described in the protocol schedule of events and consent, or inability or unwillingness to cooperate with study procedures.
5. Clinically significant abnormal safety laboratory values as determined by study physician
6. Previous history of adverse drug reaction to Levocetirizine (LTZ)
7. Unwillingness or inability to washout of medications that affect histamine response
8. Active eczema at the site where histamine laser doppler probe will be place(forearm) on the day of histamine laser doppler iontophoresis
9. Age 18 years or older at the time of enrollment.
10. Those whom are pregnant, prisoners, and/or wards of the state.
11. Currently on or has been on Tricyclic Antidepresants in past 30 days

Ages: 6 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 300 (Estimated)
Dates: Start 2021-04-28 (Actual); Primary Completion 2026-05-01 (Estimated); Study Completion 2026-05-01 (Estimated)

PRIMARY OUTCOMES:
Therapeutic response to antihistamine | 6 weeks
  Determined by change in asthma as determined by the Asthma Control Test (ACT®) or Child-Asthma Control Test (C-ACT®) based on the child's age. Asthma control will be assessed at baseline prior to randomization and then at 6 weeks during both arms (placebo and Levocetrizine) of the study.

SECONDARY OUTCOMES:
Asthma exacerbation rates | 6 weeks
  Asthma exacerbation rates will be assessed via questionnaires to assess the rate, duration, and time to first asthma exacerbation requiring systemic steroid. The investigator will also measure rates of acute office visits, emergency department/urgent care visits, and/or hospitalizations due to asthma.
  Participants will also be asked to keep a daily asthma symptom diary as a secondary measure of asthma control. Asthma control days will be defined as full calendar days without asthma symptoms, rescue medication use, or unscheduled health care visits.
  Participants will be asked to log asthma control and exacerbation data daily.
Asthma related quality of life | 6 weeks
  Quality of life will be assessed at baseline/pre-dose and at 6 weeks after each intervention arm via the validated questionnaires, Standardized Pediatric Asthma Quality of Life Questionnaire (PAQLQ(S)) and Pediatric Asthma Caregiver's Quality of Life Questionnaire (PACQLQ) to assess child and parental quality of life.

CONTACTS AND LOCATIONS:
Locations (1):
- Children's Mercy Hospital, Kansas City, Missouri, United States

IPD SHARING:
Plan to Share IPD: No